CLINICAL TRIAL: NCT06250296
Title: Evaluation of a New Recovery-oriented Model of Care on Psychiatric Inpatient Wards.
Brief Title: Evaluation of a New Recovery-oriented Model of Psychiatric Inpatient Care
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: Fondation Privée des HUG (Unknown); IF International Foundation (Unknown)
Responsible Party: Principal Investigator, Alexandre Wullschleger, MD, Principal investigator, University Hospital, Geneva
Other Study IDs: RP-07-06
Record Dates: First submitted 2024-01-29; First posted 2024-02-09 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Psychiatric Hospitalization; Coercion; Recovery
Keywords: psychiatric inpatient care; coercion; recovery; patient satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group: All patients admitted to the ward implementing the foreseen intervention as to February 2024 (pilot phase)
  Interventions: Other: New model of psychiatric inpatient care
- Control group: All patients admitted to the two wards implementing the foreseen intervention after the initial pilot phase

INTERVENTIONS:
Other: New model of psychiatric inpatient care — The intervention envisages major structural changes in wards, in particular the reorganization of clinical discussion and decision-making spaces, as well as the medical and nursing referral system, and the inclusion of relatives in care:
  * Treatment planning involving the patient, with a focus on his or her needs and resources.
  * Care by referral teams, present every day of the week, to ensure continuity and consistency of care.
  * As few decisions as possible made without the patient, and transparency in decision-making.
  * Emphasis on the subjective meaning of illness, beyond symptoms.
  * Greater visibility of care planning for patients, who will benefit from weekly agendas
  * Closer collaboration with relatives, through open invitations to all clinical discussions, telephone hotlines and meeting times.
  * Openness to the network and community care, by promoting communication and exchanges between all stakeholders, and the development of early warning tools such as the joint crisis plan.
  Groups: Intervention group

SUMMARY:
This project will study the effects of a major reorganization of psychiatric inpatient wards. This reorganization will affect many aspects of day-to-day work, with the aim of improving the individualization of care, the integration of relatives and the participation of the patients in treatment planning. This new organization will initially involve a first pilot ward, before being extended to other wards.

The aim of this project is to understand whether this new organization has positive effects on the use of coercive measures, the average length of stay, the improvement in patients' clinical condition, as well as on patient satisfaction, their perception of coercion, the wards' atmosphere on the unit and patients' personal recovery.

All patients admitted to three wards of the Division of adult psychiatry of the Geneva University Hospital aged 18 and over, with a good knowledge of French and being treated for any type of diagnosis except dementia, are invited to take part in the study. They will be assessed at discharge regarding the selected outcomes. The study will last 18 months: during the first 9 months, the new model will be applied on the pilot ward, and the wo other wards will serve as comparison wards. After 9 months, the model will also be applied to these other two wards.

DETAILED DESCRIPTION:
The project is designed as a prospective, observational study, supporting the planned reorganization of inpatient care with the implementation of a new recovery-oriented model of care. As part of this reorganization, the new model will be first implemented as a pilot on a first acute psychiatric ward. After nine months, it is planned to be generalized to two comparable other acute wards. These two wards will serve within the current project as a comparison group to assess the effects of the new model.

Patients hospitalized on these three wards will be included in the study over a period of 18 months, covering the initial implementation of the model and its subsequent extension to the other two wards.

Three psychiatric wards of the Division of adult Psychiatry (SPA) will participate in the study. These wards are dedicated to general psychiatric admissions following a sectorization plan and operate with an open-door policy, wherein the wards' doors are uninterruptedly open between 7:30 am. and 11 pm. Patients aged 18 to 65 with all types of diagnosis at the exception of primary substance-abuse disorders and dementia, which are mainly treated in other divisions, are treated on these wards.

All patients admitted to these wards during the study period will be considered for participation. All diagnoses will be included, except for dementia. Patients who are not able to give their written consent to participation and/or with insufficient knowledge of French will be excluded from the trial.

Patient fulfilling the inclusion criteria will be contacted before discharge and offered to participate in the study. They will be informed in writing of the purpose of the study and their written consent will be collected.

Data on coercive measures, length of stay as well as socio-demographic characteristics, diagnosis and admission and discharge HoNOS scores will be extracted from the patients' electronic record.

The assessment of patients' satisfaction, perceived coercion, personal recovery, patients' appraisal of the ward atmosphere, and their perception of care as supporting to their recovery will be carried at discharge using digital questionnaires on the REDCAP platform, using tablets. The planned assessment will take about 30 to 45 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in one of the three participating wards

Exclusion Criteria:

* Incapacity to give informed consent
* Insufficient knowledge of French

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the three participating wards during the study period will be considered for participation. All diagnoses will be included, except for dementia. Patients who are not able to give their written consent to participation and/or with insufficient knowledge of French will be excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Coercive measures | For each included participant at discharge from hospital, throughout the study (18 months)
  Number, type and duration of used coercive measures (seclusion or forced medication)

SECONDARY OUTCOMES:
Length of stay | For each included participant at discharge from hospital, throughout the study (18 months)
  Length of hospital stay in days
Symptom burden | For each included participant at discharge from hospital, throughout the study (18 months)
  Burden of symptoms measured at admission and discharge using the Health of Nations Outcome Scale (HoNOS). This scale comprises 12 items rated on a scale from 0 to 4. Final score between 0 and 48. Higher scores indicate higher burden of symptoms.
Length of stay under involuntary status | For each included participant at discharge from hospital, throughout the study (18 months)
  Percentage of hospital stay under involuntary status
Personal recovery | For each included participant at discharge from hospital, throughout the study (18 months)
  Level of personal recovery measured by the Recovery Assessment Scale (RAS-R). The RAS-R comprises 24 items rated on a 5-point Likert scale (1 to 5). The scale is scored by summing the responses for each of the items. total scores range from 24 to 120. Higher scores indicate better recovery.
Subjective coercion 1 | For each included participant at discharge from hospital, throughout the study (18 months)
  Level of subjective coercion measured by the Coercion Ladder (CL). The Coercion Ladder is an analog scale ranging from 1 to 10. Higher scores indicate higher levels of perceived coercion.
Subjective coercion 2 | For each included participant at discharge from hospital, throughout the study (18 months)
  Level of subjective coercion measured by the Experienced Coercion Scale (ECS). The ECS comprises 15 items rated on a 5-point Likert scale (0-4). Two items (5 and 6) are reverse scored. The average sum score is used for interpretation. Higher scores indicate higher levels of perceived coercion.
Ward atmosphere | For each included participant at discharge from hospital, throughout the study (18 months)
  Quality of the ward atmosphere measured by the Essen Climate Evaluation Schema (EssenCES). The EssenCES comprises 15 items rated on a 5-point Likert scale (0-4). Three subscores are built by adding the items scores following the scoring sheet: Patients' Cohesion, Experienced Safety, Therapeutic Hold. Higher scores indicate a better perceived atmosphere in the three dimensions.
Patients' satisfaction | For each included participant at discharge from hospital, throughout the study (18 months)
  Level of patients' satisfaction measured by the satisfaction questionnaire of the Swiss National Association for Quality Development in Hospitals and Clinics. This questionnaire comprises 6 items, each rated on a 5-Likert scale (1 to 5). The mean of each item score will be used for analysis.
Recovery-orientation of services | For each included participant at discharge from hospital, throughout the study (18 months)
  Patients' perception of the wards' level of Recovery-orientation measured by the Recovery Self-Assessment (RSA). The RSA comprises 32 items rated on a 5-point Likert scale. Total scores range from 32 to 160. Higher scores indicate a better perception of services as supporting for the recovery process.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Wullschleger, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- HUG - Hôpital de Belle-Idée, Thônex, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided